CLINICAL TRIAL: NCT01418469
Title: The Effects of Exercise on the Metabolic Fate of Branched Chain Amino Acids in Relation to Aging and Chronic Disease.
Brief Title: Disturbances in BCAA Metabolism and the Effects of Feeding and Exercise in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: European Dairy Association (EDA), Brussels (Unknown)
Responsible Party: Nicolaas EP Deutz, University of Arkansas for Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MEC 02-059.3
Record Dates: First submitted 2011-08-09; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; protein metabolism; branched-chain amino acid metabolism; exercise; protein feeding
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Caseins; Whey

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caseinate protein intake (Experimental): 18 mg protein/kg body weight caseinate and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Interventions: Dietary Supplement: Caseinate
- Whey protein isolate intake (Experimental): 18 mg protein/kg body weight whey protein isolate and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Interventions: Dietary Supplement: Whey protein isolate
- Soy protein intake (Experimental): 18 mg protein/kg body weight soy and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Interventions: Dietary Supplement: Soy
- soy+BCAA protein intake (Experimental): 18 mg protein/kg body weight soy+BCAA and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Interventions: Dietary Supplement: soy+BCAA

INTERVENTIONS:
Dietary Supplement: Caseinate — 18 mg protein/kg body weight caseinate and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Other Names: casein
  Arms: Caseinate protein intake
Dietary Supplement: Whey protein isolate — 18 mg protein/kg body weight whey protein isolate and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Other Names: Whey
  Arms: Whey protein isolate intake
Dietary Supplement: Soy — 18 mg protein/kg body weight soy and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Arms: Soy protein intake
Dietary Supplement: soy+BCAA — 18 mg protein/kg body weight soy+BCAA and 46 mg maltodextrin / kg body weight per 20 min sip feeding
  Arms: soy+BCAA protein intake

SUMMARY:
Studies on resting human muscle show that ingestion of the branched-chain amino acids (BCAA): leucine, valine and isoleucine have an anabolic effect on muscle protein metabolism. However, the effects of BCAA intake on protein metabolism during exercise are less clear. When BCAA were supplied as single amino acids, without other amino acids and/or carbohydrates, no effects were observed on protein kinetics. On the other hand, ingestion of BCAA during running appeared to reduce the catabolic effect of running on muscle protein metabolism. These experiments were all performed with mixtures of the BCAA with or without carbohydrates but not in the form of complete meals with food protein as a basis. Therefore, it is still unknown whether a protein meal, containing a substantial amount of BCAA is beneficial during exercise by inducing an anabolic effect.

Whey and Casein protein contain a substantial amount of BCAA in contrast to Soy protein. Therefore, it is hypothesized that milk-based proteins are a better and more physiological source of BCAA during exercise and will lead to more protein anabolism. Most of the available studies have been carried out in young and fit humans but there are hardly any data are available in the increasing population of the elderly. Therefore it is still unknown whether a BCAA rich protein meal can enhance the anabolic effect of exercise in older individuals.

Besides sarcopenia, a substantial part of the elderly is suffering from a chronic systemic disease such as chronic obstructive pulmonary disease (COPD). COPD represents an important health care problem. COPD is the fourth leading cause of death and will be the third leading cause worldwide in 2020. Besides the local impairment, COPD is a chronic wasting disease, associated with alterations in intermediary metabolism. Substantial disturbances have been found in BCAA (and related) metabolism in these patients at rest and during exercise. It might therefore be of clinical relevance to study the metabolic effects of BCAA rich protein meals in patients with COPD at rest and during exercise.

DETAILED DESCRIPTION:
In this study we investigate whether milk based protein sources of BCAA (casein and whey proteins) are superior to soy protein in the stimulation of protein anabolism before, during and after cycle exercise in COPD and healthy elderly and young subjects, and whether adding BCAA to soy protein will increase protein anabolism in these subjects.

To investigate Leucine, Isoleucine and Valine metabolism during and after exercise in COPD and healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Irreversible chronic airflow limitation (FEV1 <70% of predicted)
* Clinically stable condition

Exclusion Criteria:

* Oxygen supplementation
* Respiratory tract infection or exacerbation of his disease at least 4 weeks prior to the study
* Oral corticosteroids as maintenance medication
* Other concomitant metabolic disease (ie malignancy, cardiac failure, recent surgery, severe endocrine, hepatic or renal disorder)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-12; Primary Completion 2003-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change in Net whole body protein synthesis | 6 hours
  Net whole body protein synthesis during protein feeding and the response to a 20 min cycle exercise bout

SECONDARY OUTCOMES:
Change in whole body protein synthesis rate | 6 hours
  Whole body protein synthesis rate during protein feeding and the response to 20 min cycle exercise bout
Change in Leucine turnover | 6 hours
  Leucine turnover during protein feeding and the response to a 20 min cycle exercise bout
Change in Isoleucine turnover | 6 hours
  Isoleucine turnover during protein feeding and the response to a 20 min cycle exercise bout
Change in Valine turnover | 6 hours
  Valine turnover during protein feeding and the response to a 20 min cycle exercise bout
Change in plasma lactate concentration | 6 hours
  Plasma lactate during protein feeding and the response to a 20 min cycle exercise bout
Change in NH3 concentration | 6 hours
  Plasma NH3 during protein feeding and the response to a 20 min cycle exercise bout
Change in plasma amino acids concentrations | 6 hours
  Plasma amino acid concentrations during protein feeding and the response to a 20 min cycle exercise bout
Splanchnic extraction of amino acids during protein feeding | 6 hours
  Splanchnic extraction of amino acids during protein feeding and the response to a 20 min cycle exercise bout
Change in whole body protein breakdown rate | 6 hours
  Whole body protein breakdown rate during protein feeding and the response to cycle exercise

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas EP Deutz, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

REFERENCES:
- [Result] Engelen MP, Rutten EP, De Castro CL, Wouters EF, Schols AM, Deutz NE. Supplementation of soy protein with branched-chain amino acids alters protein metabolism in healthy elderly and even more in patients with chronic obstructive pulmonary disease. Am J Clin Nutr. 2007 Feb;85(2):431-9. doi: 10.1093/ajcn/85.2.431. PMID 17284740
- [Result] Engelen MP, Rutten EP, De Castro CL, Wouters EF, Schols AM, Deutz NE. Altered interorgan response to feeding in patients with chronic obstructive pulmonary disease. Am J Clin Nutr. 2005 Aug;82(2):366-72. doi: 10.1093/ajcn.82.2.366. PMID 16087980
- [Derived] Engelen MP, De Castro CL, Rutten EP, Wouters EF, Schols AM, Deutz NE. Enhanced anabolic response to milk protein sip feeding in elderly subjects with COPD is associated with a reduced splanchnic extraction of multiple amino acids. Clin Nutr. 2012 Oct;31(5):616-24. doi: 10.1016/j.clnu.2012.04.006. Epub 2012 Jun 6. PMID 22682082
- [Derived] Engelen MP, Rutten EP, De Castro CL, Wouters EF, Schols AM, Deutz NE. Casein protein results in higher prandial and exercise induced whole body protein anabolism than whey protein in chronic obstructive pulmonary disease. Metabolism. 2012 Sep;61(9):1289-300. doi: 10.1016/j.metabol.2012.03.001. Epub 2012 Apr 17. PMID 22512824